CLINICAL TRIAL: NCT04714411
Title: Real-World Efficacy and Safety Analysis of Omadacycline for the Treatment of Diabetic Foot Infections and Acute Osteomyelitis
Status: Recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 014.PHA.2020.A
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Foot Infection
MeSH Terms: interventions — omadacycline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective Cohort: A historical matched case cohort
- Prospective Cohort: Subjects will be screened daily via review of the EMR reports of inpatient admissions. Those receiving antibiotics with a notated source of skin/soft tissue infection or OM will be further reviewed to determine if the source of infection is a DFI with or without suspected or confirmed Acute osteomyelitis.
  Interventions: Drug: Omadacycline

INTERVENTIONS:
Drug: Omadacycline — Omadacycline monotgherapy
  Groups: Prospective Cohort

SUMMARY:
This will be a prospective, open-label, two-center study to assess the safety of omadacycline use in the treatment of hospitalized subjects with moderate to severe DFI with or without Acute osteomyelitis (AOM) who are at a high risk for development of CDI, AKI, and/or resistant pathogens compared to retrospective controls. Prospective enrollment will be continued until the sample size is achieved up to one year from start date (October 2020).

Secondary to slower than anticipated enrollment due to the COVID-19 pandemic and initial exclusion of AOM, following protocol amendment, patient enrollment will be continued until the sample size is achieved up to 18 months from amendment approval (anticipate April 2022 - October 2023). A historical matched case cohort (standard of care) at the two hospitals based on ICD10 codes associated with DFI [E11.(621, 622), E10.(621, 622); L97.(509, 521, 522, 523, 524, 529)], including subjects with AOM [M86.(08-09, 10, 16-19, 8X0, 8X7-8X9, 9) will be utilized for comparison.

DETAILED DESCRIPTION:
This is a year-long study with planned enrollment of 57 patients (in addition to 114 historical control patients) evaluating the use of omadacycline for treatment of diabetic foot infections (DFI). Omadacycline (Nuzyra®) is a FDA approved antibiotic for skin and skin structure infection and community-acquired pneumonia. This study is considered to be investigational because data is being collected on the use of Omadacycline for the treatment of DFI with or without AOM.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects will be eligible for inclusion if hospitalized, 18 years or older, diagnosed with type 1 or 2 diabetes, and have DFI with the additional clinical criteria as specified below:

  * Acute infection or worsening without systemic antimicrobials within the previous 14 days
  * At least one full or partial thickness-infected ulcer at or below the ankle AND
  * Purulent drainage OR
  * Two of the following:

    * Erythema
    * Local edema
    * Fluctuance
    * Induration
    * Increased local warmth
    * Fever
  * No systemic antimicrobials with current hospital admission for more than 48 hours prior to enrollment
* Inclusion will be based on

  * Empiric coverage based on organisms suspected to be caused by susceptible bacteria, if no culture identifies a specific organism; or
  * Confirmed susceptibility to omadacycline against any organism identified. Any subject in which a pathogen resistant to omadacycline is identified will be excluded from the study and antibiotics will be changed based on physician discretion.

    * First episodes of AOM at qualifying site of infection will be eligible for inclusion with any of the following criteria confirming the diagnosis:

      * Imaging (X-ray or MRI) confirmation of acute osteomyelitis
      * Pathology (bone biopsy/culture)
    * Not currently enrolled in any other clinical trial
    * Provides informed consent
    * Likely to be compliant with all study-related procedures and visits

Exclusion Criteria:

* Age less than 18 years
* Pregnant women
* Chronic osteomyelitis

  * Osteomyelitis of the same site previously treated with antibiotics
  * Documented presence of osteomyelitis more than 2 weeks prior to index admission
  * Necrotic or dead bone identified by pathology
  * Unclear chronicity of infection (if unable to determine acute osteomyelitis)
* Has any gangrenous ulcers or necrotizing fasciitis
* Has a pathogen known to be resistant to omadacycline
* Administration of additional systemic antibiotics in combination with omadacycline, not including topical routes or oral vancomycin/fidaxomicin given their local activity within the GI tract
* Contraindication or hypersensitivity to omadacycline/tetracyclines
* Unwilling or unable to participate in study-related procedures or visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult diabetic with DFI hospitalized, 18 years or older, diagnosed with type 1 or 2 diabetes, and have DFI with or without AOM
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2025-08-18 (Estimated); Study Completion 2025-08-18 (Estimated)

PRIMARY OUTCOMES:
AKI based on RIFLE criteria | Sept 2020 - Aug 2021
  Risk, injury, failure, loss and ESRD
Clostridioides difficile Infection | Sept 2020 - Aug 2021
  Frequency of Clostridioides difficile Infections while taking Omadacycline compared to other antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Crotty, PharmD, Principal Investigator — Methodist Health System
Locations (2):
- United States (2):
  - Methodist Dallas Medical Center, Dallas, Texas
  - Methodist Charlton Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Center for Health Statistics (US). Health, United States, 2016: With Chartbook on Long-term Trends in Health. Hyattsville (MD): National Center for Health Statistics (US); 2017 May. Report No.: 2017-1232. Available from http://www.ncbi.nlm.nih.gov/books/NBK453378/ PMID 28910066
- [Background] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Background] Singh N, Armstrong DG, Lipsky BA. Preventing foot ulcers in patients with diabetes. JAMA. 2005 Jan 12;293(2):217-28. doi: 10.1001/jama.293.2.217. PMID 15644549
- [Background] Prompers L, Huijberts M, Apelqvist J, Jude E, Piaggesi A, Bakker K, Edmonds M, Holstein P, Jirkovska A, Mauricio D, Tennvall GR, Reike H, Spraul M, Uccioli L, Urbancic V, Van Acker K, Van Baal J, Van Merode F, Schaper N. Optimal organization of health care in diabetic foot disease: introduction to the Eurodiale study. Int J Low Extrem Wounds. 2007 Mar;6(1):11-7. doi: 10.1177/1534734606297245. PMID 17344196
- [Background] Lazaro Martinez JL, Garcia Alvarez Y, Tardaguila-Garcia A, Garcia Morales E. Optimal management of diabetic foot osteomyelitis: challenges and solutions. Diabetes Metab Syndr Obes. 2019 Jun 21;12:947-959. doi: 10.2147/DMSO.S181198. eCollection 2019. PMID 31417295
- [Background] Johnson MJ, Shumway N, Bivins M, Bessesen MT. Outcomes of Limb-Sparing Surgery for Osteomyelitis in the Diabetic Foot: Importance of the Histopathologic Margin. Open Forum Infect Dis. 2019 Sep 10;6(10):ofz382. doi: 10.1093/ofid/ofz382. eCollection 2019 Oct. PMID 31660346
- [Background] Rice JB, Desai U, Cummings AK, Birnbaum HG, Skornicki M, Parsons NB. Burden of diabetic foot ulcers for medicare and private insurers. Diabetes Care. 2014;37(3):651-8. doi: 10.2337/dc13-2176. Epub 2013 Nov 1. PMID 24186882